IRB APPROVED AS MODIFIED May 07, 2019

#### RESEARCH SUBJECT INFORMATION AND CONSENT FORM

TITLE: A Phase II Pilot Study of Disulfiram and Copper Gluconate in

Patients with Metastatic Pancreatic Cancer and Rising CA-19-9 Levels While Receiving Abraxane-Gemcitabine or FOLFIRINOX

or Single-Agent Gemcitabine

PROTOCOL NO.: CAN-203

WIRB Protocol #20182808

**SPONSOR:** Cantex Pharmaceuticals, Inc.

**INVESTIGATOR:** Gayle S. Jameson, RN, MSN, ACNP-BC, AOCN

10510 N. 92<sup>nd</sup> Street Scottsdale, AZ 85258 United States of America

STUDY-RELATED

**PHONE NUMBER(S):** Gayle S. Jameson, RN, MSN, ACNP-BC, AOCN

480-323-1350 (24 hours)

A person who takes part in a research study is called a research or study subject. In this consent form "you" always refers to the research subject.

## **INTRODUCTION**

You are being asked to take part in a clinical trial, a type of research study. Your participation is entirely voluntary. To allow you to make an informed decision as to whether you want to take part in this research study, this document describes the purpose of the study, your rights and obligations, the procedures needed by the study, and the possible benefits and risks of participating. You should read all of this information carefully and discuss your questions and concerns with your study doctor or healthcare team. You may take home an unsigned copy of this consent form to think about or discuss your decision with your family, friends and anyone you choose. You should not join this research study until all of your questions are answered. A person who takes part in a research study is called a research or study subject. In this consent form, "you" always refers to the research subject.

Clinical trials include only people who choose to take part. Please take your time to make your decision. If you have any questions, you can ask your study doctor for more explanation about the clinical trial, this form, or your disease. This consent form may contain words that you do not understand. Please ask the study doctor or study staff to explain any words or information that you do not understand.

You are being asked to participate in a research study of an investigational drug called disulfiram-copper combination (also referred to as Dicopp®) for the treatment of metastatic adenocarcinoma of the pancreas. Disulfiram-copper combination is considered the study drug and has not been approved for the use described in this study by the Food and Drug Administration (FDA).

Things to know before deciding to take part in a research study:

- The main goal of a research study is to learn things to help patients in the future.
- The main goal of regular medical care is to help each patient.
- The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.
- Parts of this study may involve standard medical care. Standard care is the treatment normally given for a certain condition or illness.
- Other parts of this study may involve experimental (investigational) drugs or procedures that are being tested for a certain condition or illness. An investigational drug is one that has not been approved by the U.S. Food & Drug Administration (FDA).
- After reading the consent form and having a discussion with the research staff, you should know which parts of the study are experimental and which are standard medical care.
- Your medical records may become part of the research record. If that happens, your medical records may be looked at and/or copied by the Sponsor of this study and government agencies or other groups associated with the study.
- Your medical insurance may be billed for any standard medical care you receive during the research study. If your insurance company is billed then it may have access to the research records. Insurance companies may not pay for treatment that is part of a research study. Taking part in a research study could affect your current or future insurance coverage.

#### PURPOSE OF THE STUDY

The purpose of the study is to test disulfiram-copper combination, an investigational product, in patients with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of standard medical treatment with either protein-bound paclitaxel (Abraxane®)/gemcitabine (Gemzar®) or FOLFIRINOX (5FU, leucovorin, irinotecan, oxaliplatin combination regimen) and who have increased levels of the tumor marker CA 19-9 when there is no evidence from CT scans that your tumor is not responding to the therapy.

## Who can participate in this study?

Up to a total of 42 patients with metastatic adenocarcinoma of the pancreas receiving either protein-bound paclitaxel/gemcitabine or FOLFIRINOX who have increased levels of the tumor marker CA 19-9 when there is no evidence from CT scans that your tumor is not responding to the therapy are expected to participate in this study. Patients will be participate in this study at HonorHealth, and it is possible that patients may participate in this study, or a similar study, at other sites.

YOU MUST AGREE TO ABSTAIN FROM INGESTING ALCOHOLIC BEVERAGES AND ALCOHOL-CONTAINING MEDICATIONS AND PRODUCTS DURING THE TIME YOU ARE RECEIVING DISULFIRAM AND FOR AT LEAST 2 WEEKS AFTER DISCONTINUING DISULFIRAM.

Even though you may meet all the criteria for participation, it is possible that you will not be enrolled in this study.

You and your doctor will decide which chemotherapy regimen is most appropriate for your disease (either protein-bound paclitaxel/gemcitabine or FOLFIRINOX).

Protein-bound paclitaxel (also known as Abraxane) and gemcitabine will be given on the same day weeks 1, 2 and 3 followed by a week without treatment. This treatment will be repeated every 4 weeks (28 days) as per standard medical care.

FOLFIRINOX consists of oxaliplatin, irinotecan, leucovorin and 5-fluouracil given on the same day Weeks 1 (day 1) and 3 (day 15) every 4 weeks (28 days) as per standard medical care.

Protein-bound paclitaxel, gemcitabine, oxaliplatin, irinotecan, leucovorin and 5-fluorouracil are all FDA-approved drugs.

If while receiving one of these regimens, your CA 19-9 starts to rise without seeing progression in your radiographs, you will be given disulfiram-copper combination orally twice daily until you no longer respond to the treatment or the side effects determine that treatment cessation is the best course.

#### **PROCEDURES**

## **Screening Evaluation**

In the first part of the study, you will have an extensive evaluation of your medical condition. The purpose of this evaluation is to find out if you qualify for this research study. Screening procedures for this study are standard of care and include:

- Review and signing of the informed consent form before any study procedures can take place
- Complete medical history including pre-existing/current conditions, prior cancer therapy, and prior surgery
- Complete physical examination including height and weight
- Vital signs (blood pressure, pulse, respiratory rate, and temperature).
- Tumor imaging to include a computed tomography (CT) and/or magnetic resonance imaging (MRI) scan, as well as a FDG-PET scan, if required by your physician, of your chest, abdomen, pelvis, and any other part of your body will be completed. This would include a brain scan if your study doctor determines that it is necessary. If CT/MRI and FDG-PET scans were taken within 28 days prior to receiving your first dose, new scans are not necessary.
- Electrocardiogram (ECG)

- Collect blood for laboratory tests. About 3 tablespoons will be taken for the following tests:
  - o Complete blood count (CBC) with differential and platelet count
  - o Serum chemistry panel including liver and kidney function tests
  - Coagulation panel to include PTT and PT/INR
  - o CA 19-9 level
  - Serum pregnancy test (if applicable)
- Collect a urine sample for a urinalysis
- Review all medications taken within the last 30 days

If you are eligible to participate in this study, you will be assigned a unique ID that will be used to identify you while you are participating in the study.

Treatments will be administered in cycles. For the purposes of this study, each cycle will be 28 days long. During treatment with disulfiram-coper combination, you will be given a dosing diary to use to record daily when you take this investigational drug; each time you bring the investigational drug with you to the clinic, you will also need to bring the diary. The following assessments will be completed during each cycle on a specific day of the study:

### **Treatment Evaluations for Each Cycle**

Day 1 (except where noted)

- Directed physical exam
- Vital signs (blood pressure, pulse, respiratory rate, and temperature).
- Measurement of weight
- Body Surface Area (BSA) calculation prior to dosing
- Collect blood for laboratory tests. About 2 Tbsp. will be taken for the following tests:
  - o Hematology: CBC with differential and platelet count
  - o Blood chemistries (for liver and kidney function tests)
  - o CA19-9 level (prior to Day 1 for Cycle 1)
  - o Serum Pregnancy (if applicable)
- Collect a urine sample for a urinalysis
- Review any changes to your health since the last visit
- Review any changes to your medications since the last visit
- Administer anti-nausea medication before treatment
- Administer Paclitaxel Protein Bound and Gemcitabine OR
- Administer FOLFIRINOX OR
- Gemcitabine alone
- Receive disulfiram-copper combination medication and dosing diary for home use.
- Return disulfiram-copper remaining drug and drug diary (after Cycle 1)

### Day 8 and 15

- Directed physical exam Only for Cycle 1
- Vital signs (blood pressure, pulse, respiratory rate, and temperature) Only for Cycle 1
- Measurement of weight Only for Cycle 1
- Collect blood for laboratory tests (no blood collected for labs on Day 8 if you are in the FOLFIRINOX group). About 1 tablespoonful will be taken for the following tests:
  - o Hematology: CBC with differential and platelet count
  - o Blood chemistries (for liver and kidney function tests)
- Review any changes to your health since the last visit (via phone call on Day 8 if you are in the FOLFIRINOX group)
- Review any changes to your medications since the last visit (via phone call on Day 8 if you are in the FOLFIRINOX group)
- Administer anti-nausea medication before treatment
- Administer Paclitaxel Protein Bound and Gemcitabine (Days 8 and 15)
  OR
- Administer FOLFIRINOX (Day 15 only)
- Gemcitabine (Days 8 and 15)

## Day 22

- Directed physical exam Only for Cycle 1
- Vital signs (blood pressure, pulse, respiratory rate, and temperature) Only for Cycle 1
- Measurement of weight Only for Cycle 1
- Collect blood for laboratory tests. About 1 tablespoonful will be taken for the following tests: (Only for Cycle 1)
  - o Hematology: CBC with differential and platelet count
  - o Blood chemistries (for liver and kidney function tests)
- Review any changes to your health since the last visit (via phone call)
- Review any changes to your medications since the last visit (via phone call)

After Cycles 3, 6, and 9 a CT/MRI scan to evaluate disease status (using same imaging method used during your screening visit) will be completed at the end of the cycle prior to starting the next cycle. If disease progression is suspected, additional imaging and lab tests may be ordered. If your scan shows that your tumor(s) is not visible, you will be scheduled to complete a FDG-PET scan to confirm a complete response to the treatment.

An End of Study Treatment office visit will be performed when your study drug treatment ends for any reason. The End of Study Treatment evaluations include the following:

- Direct physical exam
- Vital signs (blood pressure, pulse, respiratory rate, and temperature).
- Measurement of weight
- ECG

- Collect blood for laboratory tests. About 1 tablespoonful will be taken for the following tests:
  - o Hematology: CBC with differential and platelet count
  - o Blood chemistries (for liver and kidney function tests)
  - o CA19-9 level
- Collect a urine sample for a urinalysis
- Review any changes to your health since the last visit
- Review any changes to your medications since the last visit
- · Return disulfiram-copper combination remaining drug and drug diary
- CT and/or MRI scan of your chest, abdomen, pelvis, and other regions as necessary. A brain scan may be done if necessary. If a CT scan was taken within 28 days prior to EOT, a new scan is not necessary.

Note that there may be additional blood draws throughout this study required for safety purposes; these will be considered "standard of care", for medical care and evaluation, and not for research purposes.

## **Post-Study Follow-up**

All subjects will continue to be evaluated by telephone after study completion or withdrawal. The study staff will contact you or your regular doctor by telephone every 12 weeks (or 3 months).

If after your last dose of study drugs you have ongoing side effects or other medical problems that started during the study, the study personnel might need to follow those conditions for a certain amount of time or until they reach an acceptable level.

Follow-up evaluations for side effects or other medical problems that started during the study may include the following:

- Physical exam
- Vital signs (blood pressure, pulse, respiratory rate, and temperature).
- Measurement of weight
- Collect blood for laboratory tests. About 1 tablespoonful will be taken for the following tests:
  - o Hematology: CBC with differential and platelet count
  - o Blood chemistries (for liver and kidney function tests)
  - o CA19-9 level
- Collect a urine sample for a urinalysis
- Review any changes to your health since the last visit
- Review any changes to your medications since the last visit

#### RISKS AND DISCOMFORTS

As with all investigational agents, there may be unknown risks. The study drug may not control your cancer.

You may have side effects while receiving study medication. Ask the study doctor if you have any questions about the side effects described here.

Side effects may be mild or severe and in rare cases, can be life-threatening. Some side effects may go away as soon as you stop taking the study drug. In some cases, side effects can be serious, lasting or may never go away.

The study doctor may give you medicine(s) to help lessen any side effects. Your doctor will explain how these drugs must be taken.

## **Disulfiram-Alcohol Interaction**

It is imperative that you avoid alcohol-containing products, foods, drinks and medications while on this study and for at least 2 weeks after you stop taking disulfiram.

Even small amounts of alcohol consumed while taking disulfiram can cause a severe reaction. Reactions typically begin within 10 to 30 minutes after alcohol is consumed and can last up to several hours. Reactions are typically proportional to the amounts of disulfiram and alcohol ingested (the more you take, the worse the reaction).

Moderate reactions to consuming alcohol while on disulfiram may include the following:

- Sweating
- Rapid breathing
- Difficulty breathing
- Alcoholic breath odor
- Blurred vision
- Head and neck throbbing
- Thirst
- Nausea
- Vomiting

- Vertigo (feeling off balance)
- Fainting
- Uneasiness
- Confusion
- Weakness
- Chest pain/palpitations
- Low blood pressure
- Fast heartbeat
- Warmth and flushing, particularly on upper chest and face

Severe reactions to consuming alcohol while on disulfiram may include the following:

- Slowed breathing
- Sudden loss of blood flow to the brain and other vital organs
- Irregular heartbeat
- Heart attack (in individuals with preexisting coronary artery disease)
- Seizures
- Unconsciousness
- Death
- Sudden heart failure (affecting the chambers of the heart, in individuals with preexisting myocardial dysfunction)

Disulfiram has been approved by the FDA since 1951 for the treatment of alcoholism, therefore, many people have taken it. The potential side effects listed below are based on reports from patients who have taken disulfiram in the past.

#### Serious side effects with Disulfiram:

- Alcohol intolerance
- An allergic reaction (swelling of your lips, tongue, or face; shortness of breath; closing of your throat; or hives)
- Seizures
- Extreme tiredness
- Dark urine
- Yellowing of the skin or eyes (jaundice) which can be a sign of liver damage
- Large appetite changes
- Weakness, dizziness or loss of coordination
- Hepatitis (a disease of the liver)
- Severe diarrhea or vomiting

#### Less serious side effects from disulfiram:

- Skin rash or acne
- Mild headaches
- Mild drowsiness or tiredness
- Impotence
- Metallic taste in the mouth; or swollen or sore tongue
- Increases in liver function tests

### Serious side effects with copper gluconate:

- Coma
- Diarrhea
- Stomach pain and discomfort
- Blood in urine
- Low blood pressure
- Yellowing of the skin or eyes (jaundice)
- Vomiting

## Less serious side effects from copper gluconate:

Metallic taste

#### **Common side effects of Paclitaxel Protein Bound:**

- Anemia
- Fatigue
- Hair loss (reversible)
- Joint and muscle pain
- Low white blood cell count (which may temporarily place you at risk for infection)
- Nausea
- Numbness, tingling or burning of hands and feet
- Tiredness and weakness

#### Less common side effects related to Paclitaxel Protein Bound:

- Low platelet count (which can lead to bruising or bleeding)
- Appetite loss
- Constipation
- Diarrhea
- Edema (fluid retention)
- Fever
- Irregular heartbeat
- Irritation or bruising at the site of the infusion
- Itching
- Mouth or lip sores
- Nail changes
- Vomiting

#### Rare side effects related to Paclitaxel Protein Bound:

- Allergic reaction
- Cough
- Difficulty breathing
- Congestive heart failure (the heart does not pump blood effectively)
- Left ventricular dysfunction (when a part of the heart, the left ventricle muscle, does not contract as well as it should which may lead to heart failure)
- Kidney (abnormal function or failure)
- Liver function tests abnormal
- Low blood pressure
- Pulmonary edema (fluid in lungs)
- Rash
- Visual disturbances (temporary), (flashing lights or blurry vision)

#### **Common side effects related to Gemcitabine:**

- Anemia (low red blood cell count which may cause you to feel tired, look pale, and have shortness of breath)
- Constipation
- Diarrhea
- Fever
- Flu-like symptoms (fever, feeling tired, loss of appetite, chills and cough)
- Hair loss (reversible)
- Liver function tests abnormal
- Low platelet count (which can lead to bruising or bleeding)
- Low white blood cell count (which may temporarily place you at risk for infection)
- Nausea
- Rash
- Vomiting

#### Less common side effects related to Gemcitabine:

- Edema (fluid retention)
- Fatigue
- Irritation or bruising at the site of the infusion
- Itching
- Mouth or lip sores
- Tingling, prickling of the skin

## Rare toxicities related to Gemcitabine:

- Allergic reaction
- Blood and protein in the urine
- Difficulty breathing
- Abnormal kidney function or failure
- Hemolytic uremic syndrome (abnormal clotting and kidney failure)

#### Common side effects related to 5-Fluorouracil:

- Diarrhea
- Nausea and possible occasional vomiting
- Mouth sores
- Poor appetite
- Watery eyes, sensitivity to light (photophobia)
- Taste changes, metallic taste in mouth during infusion
- Discoloration along vein through which the medication is given
- Anemia (low red blood cell count which may cause you to feel tired, look pale, and have shortness of breath)
- Low platelet count (which can lead to bruising or bleeding)
- Low white blood cell count (which may temporarily place you at risk for infection)

#### Less common side effects related to 5-Fluorouracil:

- Skin reactions: dry, cracking, peeling skin.
- Darkening of the skin (hyperpigmentation)
- Hair thinning
- Nail changes: discoloration, loss of nails (rare)
- Hand-foot syndrome (Palmar-plantar erythrodysesthesia or PPE) skin rash, swelling, redness, pain and/or peeling of the skin of the palms of hands and soles of feet

## Common side effects related to Oxaliplatin:

- Numbness and tingling and cramping of the hands or feet often triggered by cold
- Nausea and vomiting
- Diarrhea
- Mouth sores

- Anemia (low red blood cell count which may cause you to feel tired, look pale, and have shortness of breath)
- Low platelet count (which can lead to bruising or bleeding)
- Low white blood cell count (which may temporarily place you at risk for infection)
- Fatigue
- Loss of appetite

## Less common side effects related to Oxaliplatin:

- Constipation
- Fever
- Generalized pain
- Headache
- Cough
- Temporary increases in blood tests measuring liver function
- Allergic reaction

## Rare side effects related to Oxaliplatin:

• Feeling of difficulty swallowing, shortness of breath, jaw spasm, abnormal tongue sensation and feeling of chest pressure.

#### Common side effects related to Irinotecan:

- Diarrhea two types: early and late forms
- Early diarrhea: Occurring within 24 hours of receiving drug, accompanied by symptoms runny nose, increased salivation, watery eyes, sweating, flushing, abdominal cramping. (This can occur while the drug is being administered. If so, alert your healthcare professional promptly. Medication can be given to stop and/or lessen this early side effect)
- Late diarrhea: Occurring greater than 24 hours of receiving drug, usually peaks at about 11 days after treatment. Because of concerns of dehydration and electrolyte imbalances with diarrhea it is important to be in contact with health care professionals for monitoring, and for medication and diet modifications advice.
- Nausea and vomiting.
- Weakness
- Anemia (low red blood cell count which may cause you to feel tired, look pale, and have shortness of breath)
- Low white blood cell count (which may temporarily place you at risk for infection)
- Hair loss
- Poor appetite
- Fever
- Weight loss

#### Less common side effects related to Irinotecan:

- Constipation
- Shortness of breath
- Sleep problems, insomnia

- Cough
- Headache
- Dehydration
- Chills
- Skin rash
- Flatulence, gas
- Flushing of face during infusion
- Mouth sores
- Heartburn
- Swelling of feet and ankles

#### Rare side effects related to Leucovorin:

- Nausea and vomiting
- Allergic reaction rash, itching, facial flushing

## **Side Effects of palonosetron (Aloxi®):**

Palonosetron will be given by IV before the paclitaxel protein bound, cisplatin and gemcitabine to prevent nausea and vomiting that you may experience.

Less serious side effects that can occur include:

- Headache
- Constipation
- pain, redness swelling or a lump under your skin where the needle is placed

More serious side effects that can occur include:

- allergic reaction (symptoms include hives, swelling of the face or hands, trouble breathing, tingling in your mouth or throat and/or chest tightness)
- anxiety
- restlessness
- fever
- sweating
- muscle spasms
- nausea and/or vomiting
- diarrhea
- lightheadedness, dizziness, fainting
- chest pain and/or irregular heartbeat

## **Side Effects of fosaprepitant (Emend®):**

Fosaprepitant will be given by IV before the paclitaxel protein bound, cisplatin and gemcitabine to prevent nausea and vomiting. In addition, you may receive fosaprepitant orally to take on your own to prevent any nausea and vomiting that you may experience at home.

Less serious side effects that can occur include:

- nausea and/or vomiting
- heartburn
- stomach pain
- diarrhea or constipation
- loss of appetite
- hiccups
- increased thirst or hot, dry skin
- weakness, dizziness, tired feeling
- headache
- ringing in your ears
- fever, chills, body aches, flu symptoms
- sleep problems (insomnia)
- pain or a hard lump where the medicine was injected.

More serious side effects that can occur include:

- feeling light-headed
- fainting
- slow heart rate
- pale skin, easy bruising or bleeding
- pain or burning when you urinate

## **Side Effects of Dexamethasone:**

Dexamethasone will be given by IV before the paclitaxel protein bound, cisplatin and gemcitabine to prevent nausea and vomiting that you may experience.

Less serious side effects that can occur include:

- upset stomach
- stomach irritation
- vomiting
- headache
- dizziness
- insomnia
- restlessness
- depression
- anxiety
- acne
- elevated blood sugars
- increased hair growth
- easy bruising
- irregular or absent menstrual periods

More serious side effects that can occur include:

- skin rash
- swollen face, lower legs, or ankles
- vision problems
- cold or infection that lasts a long time
- muscle weakness
- black or tarry stool

## Side Effects of ondansetron (Zofran®):

Ondansetron may be given in lieu or in addition to fosaprepitant to prevent/treat nausea and vomiting. Your doctor will decide what the best course of treatment is to prevent/treat any nausea/vomiting that you may experience.

Less serious side effects that can occur include:

- headache
- constipation
- weakness
- tiredness
- chills
- drowsiness

More serious side effects that can occur include:

- blurred vision or vision loss
- rash
- hives
- itching
- swelling of the eyes, face, lips, tongue, throat, hands, feet, ankles, or lower legs
- hoarseness
- difficulty breathing or swallowing
- chest pain
- shortness of breath
- dizziness, light-headedness, or fainting
- fast, slow or irregular heartbeat
- agitation
- hallucinations (seeing things or hearing voices that do not exist)
- fever
- excessive sweating
- confusion
- nausea, vomiting, or diarrhea
- loss of coordination
- stiff or twitching muscles
- seizures
- coma (loss of consciousness)

Additional medications not listed may be given to help treat any side effects. Please talk to your study doctor regarding any questions or concerns you may have about any side effects you are experiencing.

## Reproductive risks

Women of childbearing potential are women who are biologically capable of becoming pregnant. This includes women who are using contraceptives or whose sexual partner is either sterile or using contraceptives.

The study drugs may affect an unborn child or nursing infant. The risks to an unborn child or nursing infant are not fully known. These drugs may also cause changes to eggs in women.

The following information is for women who are able to become pregnant:

- It is important that you do not become pregnant while in this study. If you become pregnant, you will be taken off this study.
- You must have a negative serum (blood) pregnancy test before you start taking the study drugs.
- If you do become pregnant or suspect you are pregnant, while you are on this study or within 30 days after the last dose of study treatment, you must notify your study doctor immediately.
- You must not breast feed at any time you are in this study since any drugs you are taking may also affect the child.

## **Birth Control Requirements for Female Participants:**

If you are sexually active and able to become pregnant, you must agree to use two forms of highly effective birth control methods listed below:

- Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
- Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- Intrauterine device (IUD)
- Abstinence (no sex)

# NOTE: Hormonal contraceptives alone are not considered an acceptable method of birth control for this study.

You must use birth control for the entire study and for at least 30 days after your last dose of study treatment.

## **Birth Control Requirements for Male Participants:**

The study drugs may have a harmful effect on sperm. This can lead to damage to a fetus or embryo (developing unborn baby). If you are a fertile male, you must not impregnate a female while in this study.

If you are sexually active, and able to father a child, you must agree to use two forms of birth control methods listed below:

- Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- Hormonal methods used by your partner, such as birth control pills, patches, injections, vaginal ring, or implants
- Intrauterine device (IUD) used by your partner
- Abstinence (no sex)

## **Risks from Study Procedures:**

- **Risk of Infection:** Subjects that develop a fever should notify their study doctor or the study team as soon as possible and may be asked to return to the study location for evaluation and possible treatment. If you develop a fever, you should begin taking the antibiotic provided to you at the first visit immediately. We will take reasonable safeguards to minimize known and potential risks but unknown and/or unanticipated side effects might occur. Some side effects go away when the study drugs are stopped. Others may be long lasting.
- Risks with Intravenous (IV) Drug Administration: Temporary irritation and bruising may occur at the infusion site. There may also be discomfort, pain, or bruising from the needle puncture. In rare cases, an infection may also occur at the site of the needle stick.
- Risks of a Blood Draw: Risks can also occur during blood draws. The risk of blood drawing may include bleeding, pain, lightheadedness, fainting, bruising, clotting, discomfort, and/or infection at the site of the needle stick. Your blood will be drawn weekly during the study. Depending on your condition, your study doctor may wish to perform additional blood draws.
- **Electrocardiogram** (**ECG**): This test uses small sticky pads that are placed on your chest and limbs to measure the electrical activity of your heart. There may be mild discomfort from the sticky pads and a possibility of the skin being irritated by the adhesive on the sticky pads. Chest hair may need to be shaved prior to the placement of the sticky pads.
- CT (computed tomography) scans: You may experience fear of being in a narrow or enclosed space while having a CT/MRI scan. You will be asked not to move during the test and to relax and breathe normally. A CT scan exposes you to a small dose of radiation. Although all radiation you receive builds up over your lifetime, this amount of radiation should not create a significant risk to your health. Contrast dye is usually injected when you get a CT scan. The contrast dye may cause pain or burning when it is injected, and may worsen kidney function in patients who already have kidney disease or who are dehydrated (have not had enough liquids that day). The contrast dye may also cause an allergic reaction, which could be severe and life-threatening.
- MRI (magnetic resonance imaging): There are risks from an MRI if you are pregnant or have one of the following: an artificial heart valve, pacemaker, metal plate, pin, or other metallic objects in your body (including gun shot or shrapnel). You may also become anxious from lying in a tight space without moving. The MRI scan does not cause any pain and does not expose you to x-ray radiation.

• **PET** (positron emission tomography) scan: A PET scan is an imaging technique that uses positively charged particles (radioactive positrons) to detect subtle changes in the body's metabolism and chemical activities. A PET scan provides a color-coded image of the body's function, rather than its structure. You may experience a mild skin prick when a substance called a tracer is injected into the vein. The tracer is radioactive but short lived and poses little to no risk.

You must use birth control for the entire study and for at least 30 days after your last dose of study drug. If your partner becomes pregnant while you are on the study or within 30 days of receiving the last dose of study medication, you will need to report this to your study doctor.

#### **Other Risks**

There may be side effects that are not known at this time. Your condition may not get better or may get worse during this study. The dose you receive may be too low to have the best effect, or so high that it causes bad side effects.

Only you should take the study drug. It must be kept out of the reach of children or anyone else who may not be able to read or understand the label.

#### **NEW INFORMATION**

You will be told about anything new that might change your decision to be in this study. If there is new information, you may be asked to sign a new consent form.

#### **BENEFITS**

It cannot be promised that you will receive any medical benefits from being in this study.

There may be no direct medical benefit to you from participating in this study, except you may gain information about your health from the different tests that are done as part of the study. Information obtained from this study will benefit the Sponsor. It might also lead to treatments that help others in the future.

#### **COSTS**

Honor Health will pay for all procedures and tests done specifically for this research study. Those treatments, procedures (including drug infusions) and tests that you would be likely to receive whether you were in the study or not, are not paid for by the study Sponsor, and are considered "standard of care" for your medical condition. If you have health insurance, the cost of these "standard of care" services will be billed to your insurance company. Your health insurance may not cover these costs because of your participation in this research study. If it does not, the costs will be your responsibility. If you do not have health insurance, the cost of these "standard of care" services will be billed to you.

You might have unexpected expenses from being in this study. Ask your Patient Financial Counselor to discuss the costs that will or will not be covered by the Sponsor. This discussion should include who will pay the costs of treating possible side effects.

You may need to receive medical care that is not listed in this document. HonorHealth will not cover the costs of that care.

You may want to talk with your insurance company about its payment policy for standard medical care given during a research study. If your insurance company does not pay, you may be billed for those charges.

#### PAYMENT FOR PARTICIPATION

You will be paid a \$25 stipend at Screening, Day 1 of each cycle, End of Treatment and Follow-up visits.

#### ALTERNATIVE TREATMENT

There are other treatment options for locally advanced pancreatic cancer. These options include other chemotherapy regimens, radiation, or other experimental therapy. Your study doctor will explain the other options available to you. You do not have to participate in this study to receive treatment for your condition. You may also choose to receive no treatment for your cancer.

If you decide that you don't want any more active treatment, one of your options is called "comfort care." Comfort care includes pain medication and other support. It aims to maintain your comfort and dignity rather than cure disease. Usually this care can be provided at home.

If you think you might prefer comfort care, please discuss this with your family, friends and your doctor.

## CONFIDENTIALITY OF YOUR INFORMATION COLLECTED DURING THE STUDY

As required by the Federal Health Insurance Portability and Accountability Act (HIPAA), every effort will be made to safeguard the confidentiality of information that identifies you and relates to your past, present and future physical and mental health. We will do our best to make sure that the personal information obtained during the course of this research study will be kept private However, we cannot guarantee total privacy. Your personal information may be given out if required by law.

Unless required by law, you will not be identified on any electronic form by name, social security number, address and telephone number or any other information that can directly identify you. The information shared with the sponsor is protected by the use of a code, which is a number specifically assigned to you. The study doctor is in control of the code needed to connect your data to you, but the study doctor will not send the list with the code to the sponsor. However, the study forms may contain other information about you, such as your age, sex and medical history. It is possible that this other information could be used to identify you even though your name does not appear.

The results of this study may be published by the sponsor, including in a medical journal and shown at medical meetings. You will not be identified (by name or any other means, e.g., photo) in any of these publications.

Because this research is regulated by the Food and Drug Administration (FDA), the FDA may inspect records related to this research, which may include your protected health information or other information about you derived or maintained as part of this study.

Information derived from this study may be used for research purposes that may include publication and teaching. However, information used for publication and teaching will not disclose your identity.

#### **COMPENSATION FOR INJURY**

We will make every effort to prevent study-related injuries and illness. If you are injured or become ill while you are in the study and the illness or injury is due to your participation in this study, you may go to any emergency room or urgent care facility to seek medical treatment. If it is determined that the injury or illness is not related to the research, the costs of this care may be charged to you or to your health insurer. No funds are available from HonorHealth to compensate you for a study-related injury or illness. This does not mean that you are giving up any of your legal rights.

The study doctor will provide you medical care if you need it, and will also treat you for any complications that may occur during your participation in the study. If you become ill or are injured as a direct result of your participation in this study, you will be provided the reasonable and necessary treatment for that injury or illness. The bills for the injury or illness not caused by study participation may be billed to your medical insurance or to your third party or governmental programs in which you participate.

The Sponsor, Cantex Pharmaceuticals, Inc., will reimburse you for any reasonable, necessary medical expenses, including hospitalization that you incur as a direct result of receiving Disulfiram-Copper combination as written in the protocol. Expense reimbursement will be determined by the Sponsor and your study doctor. The Sponsor will not provide reimbursements for injuries, illnesses, or conditions that (1) are unrelated to Disulfiram-Copper combination; (2) are related to Abraxane-Gemcitabine or FOLFIRINOX; (3) are related to the natural course of any underlying disease or treatment; (4) existed prior to Disulfiram-Copper combination administered to you on the study; or (5) related to the intake of alcohol in conjunction with disulfiram, as prohibited by the study protocol. No funds have been set aside to provide you with any other form of compensation, such as reimbursement for lost wages.

#### **VOLUNTARY PARTICIPATION AND WITHDRAWAL**

Your participation in this study is voluntary. You may decide not to take part or you may leave the study at any time. Your decision will not cause any penalty or loss of benefits to which you are entitled.

Your participation in this study may be stopped at any time by the study doctor or the Sponsor without your consent for any of the following reasons:

- vour cancer becomes worse
- side effects arise which prevent further study treatment
- you decide to withdraw from the study

- changes in your condition occur that lead your study doctor to believe that it would be harmful for you to receive further study treatment
- you become pregnant or fail to use adequate birth control (if you are of child-bearing potential)
- another anticancer medication is started
- you cannot or will not follow the instructions for participation in the study
- the study doctor decides it is in your best interest not to continue in the study.

If you leave the study before the planned final visit, you may be asked by the study doctor to have some tests or procedures done so that you leave the study safely.

#### SOURCE OF FUNDING FOR THE STUDY

HonorHealth has received funding from the Translational Genomics (TGen) Foundation to conduct this research study. Your study doctor is receiving a salary from HonorHealth as an employee but will not receive any additional payments for conducting this study.

## AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

## What information will be collected by the study doctor and his research staff for this study?

The study doctor will collect your personal and medical information. This may include:

- Past and present medical records,
- Research records,
- Records about phone calls made as part of this research,
- Records about your study visits.

## Who may use and give out information about you?

The study doctor and his research staff conducting the research.

### Who will receive your personal and medical information collected?

Information from this study will be given to the study Sponsor. "Sponsor" is the person or entity that initiates, provides oversight of activities within the study, and includes any persons or companies that are contracted by the Sponsor to have access to the research information during and after the study. Medical records which identify you and the consent form signed by you will be looked at and collected for research purposes by:

- Cantex Pharmaceuticals, the Sponsor,
- HonorHealth Research Institute, the study site
- Translational Genomics (TGen) Foundation, providing funding for the study.

## Your information may be given to:

- The U.S. Food and Drug Administration (FDA),
- Department of Health and Human Services (DHHS) agencies,
- Governmental agencies in other countries,

- Governmental agencies to whom certain diseases (reportable diseases) must be reported,
- Western Institutional Review Board (WIRB®),
- HonorHealth Institutional Review Board.

The HonorHealth IRB and the HonorHealth Research Institute have the authority to review and monitor all records related to this research.

## Why will this information be used and/or given to others?

- for research purposes as described in this consent form,
- for consideration by the FDA or any governmental agencies in other countries for drug approval,
- to ensure the study was conducted as approved by the FDA and IRB,
- to be used for future research purposes.

## What will happen if you decide not to give permission to use and give out your private health information?

You cannot be in this research study.

## Will you have access to the information collected during the study?

To maintain the integrity of this research study, you will not have access to your personal health information related to this research until the study is complete. At the conclusion of the research and at your request, you may request access to your health information that HonorHealth maintains in a designated record set, which means a set of data that includes medical information or billing records used in whole or in part by your doctors or other health care providers at HonorHealth. If it is necessary for your care, your health information will be provided to you or your physician.

## Does this authorization expire?

This authorization does not expire unless it is canceled by you in writing.

#### Can this authorization be withdrawn or canceled?

You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the study doctor. If you withdraw your permission, you will not be able to stay in this study.

When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

## Is my health information protected after it has been given to others?

There is a risk that your information will be given to others without your permission. Absolute confidentiality cannot be guaranteed because of the need to give information to these parties.

## **QUESTIONS**

Contact Gayle S. Jameson, RN, MSN, ACNP-BC, AOCN at 480-323-1350 (24 hours) for any of the following reasons:

- if you have any questions about your participation in this study,
- if at any time you feel you have had a research-related injury or a reaction to the study drug, or
- if you have questions, concerns, or complaints about the research.

If you have questions about your rights as a research subject or if you have questions, concerns, input, or complaints about the research, you may contact:

Western Institutional Review Board® (WIRB®) 1019 39<sup>th</sup> Avenue SE, Suite 120 Puyallup, Washington 98374 Telephone: 1-800-562-4789 or 360-252-2500

E-mail: Help@wirb.com

WIRB is a group of people who independently review research.

WIRB will not be able to answer some study-specific questions, such as questions about appointment times. However, you may contact WIRB if the research staff cannot be reached or if you wish to talk to someone other than the research staff.

Do not sign this consent form unless you have had a chance to ask questions and have gotten satisfactory answers.

If you agree to be in this study, you will receive a signed and dated copy of this consent form for your records.

## ClinicalTrials.gov

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

IRB APPROVED AS MODIFIED May 07, 2019

#### **CONSENT**

I have read this consent form and understand what has been discussed. All my questions about the study and my part in it have been answered. I voluntarily consent to be in this research study.

I authorize the use and disclosure of my health information to the parties listed in the authorization section of this consent for the purposes described above.

| By signing this consent form, I have not given up an | y of my legal rights. |
|---|---|
| Subject Name (printed) | |
| Signature of Subject | Date |
| Name of Person Conducting Informed Consent Discussion (printed) | |
| Signature of Person Conducting Informed Consent Discussion | Date |
| Use this witness section only if applicable | |
| If this consent form is read to the subject becau<br>impartial witness not affiliated with the research of<br>and sign the following statement: | |
| I confirm that the information in the consent faccurately explained to, and apparently understood to be in the research study. | |
| Signature of Impartial Witness | Date |

Note: This signature block cannot be used for translations into another language. A translated consent form is necessary for enrolling subjects who do not speak English.